CLINICAL TRIAL: NCT05939999
Title: Effects of Elastic Tape on Pulmonary Rehabilitation of Patients with Chronic Obstructive Pulmonary Disease
Acronym: ETReaCOPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/09628-1
Record Dates: First submitted 2023-06-29; First posted 2023-07-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: rehabilitation; exercise capacity; health-related quality of life; elastic tape
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluations will be conducted blindly, that is, by an evaluator who will not be directly involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elastic tape (ET) (Experimental): The group that will participate in the 8 weeks pulmonary rehabilitation protocol using the elastic tape.
  Interventions: Other: Experimental: Elastic tape (ET)
- Sham (SH) (Sham Comparator): The group that will participate in the pulmonary rehabilitation protocol using micropore tape.
  Interventions: Other: Sham Comparator: Sham (SH)

INTERVENTIONS:
Other: Experimental: Elastic tape (ET) — The elastic tape will be allocated in the chest wall and abdomen of individuals and will be used during the 8 weeks of rehabilitation protocol.
  Arms: Elastic tape (ET)
Other: Sham Comparator: Sham (SH) — The micropore tape will be allocated in the chest wall and abdomen of individuals and will be used during the 8 weeks of rehabilitation protocol.
  Arms: Sham (SH)

SUMMARY:
Evaluate the effect of the use of elastic tape in chest wall and abdomen in the physical capacity, psychosocial distress levels, quality of life and anxiety, and depression symptoms of individuals with moderate to very severe chronic obstructive pulmonary disease (COPD) undergoing pulmonary rehabilitation.

DETAILED DESCRIPTION:
Individuals will be evaluated on two non-consecutive days (7 days apart). On the first visit, wil be obtained: clinical and anthropometric data and assessed clinical control [COPD Assessment Test™(CAT)], health-related quality of life [Chronic Respiratory Questionnaire (CRQ)], and anxiety and depression levels [Hospital Anxiety and Depression Scale (HADS)]. Patients will also perform a complete pulmonary function test. After, the volunteers will receive a triaxial accelerometer to assess their physical activity level (PAL) and will be instructed to return after seven days. On the second visit, patients will undergo the Incremental Shuttle Walking Test (ISWT), and the Endurance Shuttle Walking Test (ESWT), without ET.

After the assessments, the individuals will be randomized. Randomization will be computer generated (www.randomization.com) by an investigator who will not be involved in individual recruitment, evaluation, or intervention. The allocation of individuals will be secret using consecutive numbered, sealed, and opaque envelopes (concealed allocation). Initial and post-intervention assessments will be performed by an investigator who will not be involved in the recruitment, evaluation, or intervention. After inclusion, individuals will start a pulmonary rehabilitation (PR) program for eight weeks; twice a week, individuals in the ET group will have the tape applied at the beginning of each session and removed at the end. After completing the 8-week PR period, individuals will undergo the same tests performed in two visits.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to very severe COPD diagnosis according to Global Iniciative for Chronic Obstructive Lung Disease (GOLD) 2020
* Clinical stability (i.e., no exacerbations for at least 30 days)
* Male
* Non-obese (BMI ≤29.9 kg/m2)
* No musculoskeletal limitation
* Not included in a pulmonary rehabilitation program in the last 6 months.
* Do not perform home oxygen therapy

Exclusion Criteria:

* Present osteoarticular, cognitive, neurological, and/or cardiological dysfunctions that prevent physical training

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Functional Exercise Capacity: The total time reached in the Endurance Shuttle Walking Test (ESWT) | Change from baseline at 8 weeks of intervention.
  The patients will be instructed to walk in a 10-meter corridor limited by cones (with a distance of 9 meters between them), and the speed will be determined by a sound signal issued by cell phone, in this case, the speed will be determined using 85% of the maximum speed reached in the Incremental Shuttle Walking Test (ISWT) and will be constant throughout the test.

SECONDARY OUTCOMES:
Clinical Control: COPD Assessment Test™ (CAT) is a specific questionnaire for COPD that assesses the impact of the symptoms of the disease | Change from baseline at 8 weeks of intervention.
  It consists of eight items related to the health condition and is applied and validated worldwide in several langes. The maximum test score is 40 points, and the questions cover follow symptoms: cough, phlegm production, chest pressure, shortness of breath, activities of daily living, psychological aspects, sleep, and mood. Each question has six options (0-5), and the lower the score, the better the health condition.
Symptoms of Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS): The questionnaire was developed to identify symptoms of anxiety and depressive mood. | Change from baseline at 8 weeks of intervention.
  It consists of 14 multiple-choice questions divided into two subscales: anxiety (HADS-A) and depression (HADS-D), with seven questions each. The domains are categorized by the severity of the stress present: 0-7 - none; 8-10 - likely; >11 - present.
Health-related Quality of Life: was assessed by using the Chronic Respiratory Questionnaire (CRQ) | Change from baseline at 8 weeks of intervention.
  This questionnaire consists of 20 questions, divided into four domains: Fatigue (4 questions), Emotional Function (7 questions), and Self-control (4 questions) evaluated using a Likert scale with seven alternatives ranging from "never" to "always." The dyspnea domain (5 questions) has an individualized assessment in which the individual chooses from a list of 26 daily activities which are the five activities that most cause dyspnea and then grades each one again using a Likert scale with seven alternatives ranging from "unbearable shortness of breath" to "No shortness of breath." Results are expressed as the average score for each domain and the total score, and higher scores indicate a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No